CLINICAL TRIAL: NCT06908057
Title: Access to Clinical Care, Education and Screening for Underserved Children and Adults With Type 1 Diabetes (ACCESS-T1D)
Brief Title: Accessing Care, Clinical Trials and Screening for Underserved Children and Adults With Type 1 Diabetes (ACCESS-T1D)
Acronym: ACCESS-T1D
Status: Recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2130661
Record Dates: First submitted 2025-03-12; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes; Celiac Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Celiac Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood Draw — We will draw blood to measure islet-related autoantibodies and celiac disease markers with a combined research method, blood sugar, C-peptide (an indicator of insulin production that controls sugar levels) and hemoglobin A1c. Additional blood will be collected for the study of biomarkers of T1D and for long-term storage for potential future use.

SUMMARY:
The purpose of this study is to identify people with T1D or celiac disease (CD) early in the course of their disease and to improve the methods of screening for these diseases.

DETAILED DESCRIPTION:
The study will screen people who may be at risk for T1D because they have at least one person in the family with probable T1D. It can be a parent or a sibling. It can also be a second-degree relative, like nieces, nephews, aunts, uncles, grandchildren, or cousins. A relative of someone with T1D is at a higher risk of getting the disease as they are people with other autoimmune diseases. It is possible to detect T1D or CD before it shows any symptoms of high blood sugar. Sometimes, particularly in people who develop T1D in adult life, the disease is misdiagnosed as type 2 diabetes. The treatment and care for the two diseases are different.

ELIGIBILITY:
Inclusion Criteria

1. Able to provide informed consent (adults 18 and above) and assent if seven or above. Legally authorized representative (LAR) is able to provide consent in case of minors or in case of adults unable to consent.
2. Children > 2 years and adults at elevated risk of developing (or having misdiagnosed) clinically evident Stage 3 T1D because they have at least one of the following:

   i. have one or more first- or second-degree family members (siblings, parents, cousins, aunts/uncles, grandparents) diagnosed with type 1 diabetes or ii. have other autoimmune diseases such as but not limited to celiac disease, Multiple sclerosis, rheumatoid arthritis or, thyroid disease or iii. Those diagnosed with other forms of diabetes which are suspected of being T1D because of a BMI ≤28 or progression to insulin dependence within 3 years from diagnosis.
3. Resides in the following Counties: Orange, Seminole, Osceola, Lake, Volusia, Brevard, Polk, Hillsborough.

Exclusion Criteria

1. People with a diagnosis of type stage 3T1D or T1D clinical definition per ADA Standards of Care
2. History of organ transplant
3. Be deemed unable or unlikely to comply with the protocol.
4. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete study visit/s.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The targeted study population is categorized as vulnerable.
  Cognitively Impaired Adults: Cognitively impaired adults will be evaluated case to case. For example, a high functioning person with Trisomy 21 (Down's syndrome) could be a possible participant, since they are at high risk of diabetes.
  Children: above the age of two with a sibling, parent, or other first or second-degree relatives with T1D or children with another other autoimmune diseases will be able to participate. Participation involves minimal risk (not greater than that encountered for clinical purposes) with the prospect of individual benefit.
  Pregnant Women: Participation involves minimal risk (not greater than that encountered for clinical purposes) with the prospect of individual benefit.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Blood sample will be drawn for islet-related autoantibodies | Visit 1 (1 day, 1-2 hours)- Only visit for the entire study.
  A blood sample will be drawn for islet-related autoantibodies. The initial autoantibody measurement will be done with the ECL research method which detects multiple autoantibodies at once. Positive results will be confirmed with a RBA validated for clinical use.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Casu, MD, Principal Investigator — Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States